CLINICAL TRIAL: NCT00005955
Title: Phase II Treatment of Children With Newly Diagnosed Malignant Central Nervous System Tumors With Temozolomide Prior to Radiation Therapy
Brief Title: Temozolomide Followed by Radiation Therapy in Treating Children With Newly Diagnosed Malignant CNS Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Henry Friedman, MD, Duke UMC
Purpose: Treatment
Other Study IDs: 0931; DUMC-0931-02-6R3; DUMC-000931-00-5R1; DUMC-0831-99-5; NCI-G00-1799; DUMC-000931-01-6R1; CDR0000067936 (Other: NCI)
Record Dates: First submitted 2000-07-05; First posted 2003-01-27 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2009-10

CONDITIONS: Brain and Central Nervous System Tumors; Neuroblastoma
Keywords: childhood infratentorial ependymoma; childhood low-grade cerebral astrocytoma; childhood supratentorial ependymoma; childhood craniopharyngioma; localized resectable neuroblastoma; regional neuroblastoma; disseminated neuroblastoma; stage 4S neuroblastoma; childhood high-grade cerebral astrocytoma; childhood oligodendroglioma; childhood choroid plexus tumor; childhood grade I meningioma; childhood grade II meningioma; childhood grade III meningioma; untreated childhood supratentorial primitive neuroectodermal tumor; untreated childhood cerebellar astrocytoma; untreated childhood medulloblastoma; untreated childhood visual pathway and hypothalamic glioma; newly diagnosed childhood ependymoma; childhood central nervous system choriocarcinoma; childhood central nervous system embryonal tumor; childhood central nervous system mixed germ cell tumor; childhood central nervous system teratoma; childhood central nervous system yolk sac tumor
MeSH Terms: conditions — Central Nervous System Neoplasms; Neuroblastoma; Astrocytoma; Oligodendroglioma; Choroid Plexus Neoplasms | interventions — Temozolomide

INTERVENTIONS:
Drug: temozolomide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Chemotherapy combined with radiation therapy may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of temozolomide followed by radiation therapy in treating children who have newly diagnosed malignant central nervous system tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate to treatment with temozolomide in children with newly diagnosed malignant central nervous system tumors.
* Determine the toxicity of this treatment in these patients.
* Determine the overall survival in these patients for 18 months following the study after receiving this treatment.

OUTLINE: Patients are stratified according to type of disease (ependymoma vs brain stem glioma vs malignant glioma vs other).

Patients receive oral temozolomide on days 1-5. Treatment repeats every 28 days for a maximum of 4 courses in the absence of disease progression or unacceptable toxicity. Patients with a partial or complete response may receive an additional 8 courses of temozolomide following radiotherapy.

PROJECTED ACCRUAL: A maximum of 100 patients (25 per stratum) will be accrued for this study over 24-36 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed newly diagnosed malignant central nervous system tumor not requiring immediate radiotherapy
* Patients with diffuse pontine tumors do not require histological confirmation
* Eligible types include the following:

  * Ependymoma
  * Malignant glioma

    * Anaplastic astrocytoma
    * Glioblastoma multiforme
    * Anaplastic oligodendroglioma
    * Gliosarcoma
    * Anaplastic mixed oligoastrocytoma
  * Brainstem glioma
  * Primitive neuroectodermal tumor
  * Nongerminoma germ cell tumor
* At least one bidimensionally measurable lesion

  * At least 1.5 cm2 within 72 hours of surgical resection or greater than 14 days after surgery
  * Diffuse pontine tumors are not required to be measurable
* Neurologically stable

PATIENT CHARACTERISTICS:

Age:

* 4 to 21

Performance status:

* Karnofsky or Lansky 70-100%

Life expectancy:

* Greater than 12 weeks

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10 g/dL

Hepatic:

* Bilirubin less than 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase less than 2 times ULN
* SGOT and SGPT less than 2.5 times ULN

Renal:

* BUN and creatinine less than 1.5 times ULN

Other:

* Must be able to swallow capsules
* No acute infection treated with intravenous antibiotics
* No nonmalignant systemic disease that makes patient a poor medical risk
* No frequent vomiting or medical condition that may interfere with oral medication intake (e.g., partial bowel obstruction)
* No other prior or concurrent malignancies except surgically cured carcinoma in situ of the cervix or basal or squamous cell carcinoma of the skin
* HIV negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No more than one prior biologic therapy regimen
* No concurrent biologic therapy
* No concurrent growth factors or epoetin alfa

Chemotherapy:

* No more than one prior chemotherapy regimen
* No other concurrent chemotherapy

Endocrine therapy:

* No increasing doses of steroids within one week of study

Radiotherapy:

* See Disease Characteristics
* No concurrent radiotherapy

Surgery:

* At least 2 weeks, but no greater than 4 weeks, since prior surgical resection and recovered

Other:

* No other concurrent investigational drugs

Ages: 4 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 2000-08; Study Completion 2002-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry S. Friedman, MD, Study Chair — Duke University
Locations (1):
- Duke Comprehensive Cancer Center, Durham, North Carolina, United States